CLINICAL TRIAL: NCT02830009
Title: IDENTIFICATION OF A MULTI-ANALYTE PROFILE FOR PRIMARY HYPEROXALURIA AND COMPARISON WITH HEALTHY SIBLINGS AND IDIOPATHIC HYPERCALCIURIA
Acronym: PH1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-604
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Primary Hyperoxaluria Type 1; Idiopathic Hypercalciuria
MeSH Terms: conditions — Primary hyperoxaluria type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Primary Hyperoxaluria patient (Other)
  Interventions: Other: Urines samples; Other: Blood sample
- Primary Hyperoxaluria patient's siblings (Other)
  Interventions: Other: Urines samples; Other: Blood sample
- Idiopathic hypercalciuria patients (Other)
  Interventions: Other: Urines samples; Other: Blood sample
- Healthy volunteers (Other)
  Interventions: Other: Urines samples; Other: Blood sample

INTERVENTIONS:
Other: Urines samples — 24-hour urines will be collected
Other: Blood sample

SUMMARY:
The aim of this study is to know the difference between protein profiles (multi-analyte profile) of PH1 patients, idiopathic hypercalciuria (IH) patients and PH1 patients 'siblings. Idiopathic hypercalciuria is a less severe kidney disease that PH1, which also leads to the formation of kidney stones.

The aim is to identify patterns of discriminating markers associated with primary hyperoxaluria type 1 (PH1) that will significantly improve clinical diagnosis and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary hyperoxaluria, type 1 (PH1-Cohort A); OR
* Confirmed with AGXT mutation analysis (PH1-Cohort A)
* Diagnosed with idiopathic hypercalciuria (IHC- Cohort B);
* Potential subject diagnosed with PH1 or IH and has both data entered into the registry and has matched, archived random and 24-hour urine specimens obtained prior to any treatment intervention OR is consented and enrolled into the registry or this specific study during the program;
* Healthy siblings of PH1 patients known not to have PH or any another stone disease or chronic disease will be consented and enrolled into this study through the local sites where their sibling is being treated for PH1 (this study meets the criteria for expedited review through local or central IRBs);
* Healthy non-sibling controls known not to have PH or any another stone disease or chronic disease (Healthy Control-Cohort C);
* There is no upper or lower limit to the pediatric age range of enrolling infant, children and adolescent subjects, although it is understood that accurate and complete 24-hour urine collection in very young children and infants will be problematic and will be seriously considered in advance of individual patient or healthy controls enrollment;
* eGFR (Glomerular Filtration Rate) > 60 mL/min x 1.73 m2 with PH1 and IH patient cohorts matched by mean eGFR from their initial study (or registry) enrollment/ data collection.

Exclusion Criteria:

* Unwilling to provide written parent consent or adolescent assent to enroll into the International Registry or this study;
* Potential PH1, hypercalciuria, or siblings of PH1 patients with other chronic or acute illness or disease that could potentially confound proteomic results;
* Healthy intra-familial siblings unwilling to provide a blood sample for serum creatinine;
* Unwilling to provide urine specimens or permit data abstraction for the registry or this study.
* Not covered by, or having the right to, Social Security

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
presence of protein markers in urine | 24 hours

SECONDARY OUTCOMES:
Presence of discriminative and robust protein markers in urine | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon/bron, France

IPD SHARING:
Plan to Share IPD: No